CLINICAL TRIAL: NCT03655704
Title: Apabetalone for Pulmonary Arterial Hypertension: a Pilot Study
Acronym: APPRoAcH-p
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Steeve Provencher (Other)
Collaborators: Resverlogix Corp (Industry)
Responsible Party: Sponsor-Investigator, Steeve Provencher, Professor, Laval University
Organization: Laval University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CER-21723
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Apabetalone; Bromodomain-Containing Protein 4 (BRD4); BRD4 inhibitor; Feasibility pilot study; Phase 2 clinical trial; Open-label; Two-centre
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — apabetalone; MZ1 compound

STUDY DESIGN:
Intervention Model Description: Pilot study to assess the feasibility of a Phase 2 clinical trial assessing apabetalone in 10 PAH patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apabetalone (Experimental): 100mg BID for 16 weeks.
  Interventions: Drug: Apabetalone

INTERVENTIONS:
Drug: Apabetalone — A 4-week pre-treatment phase will allow ensuring that patients are on stable doses of medication. Patients will be given doses of apabetalone 100mg BID for 16 weeks. Patients will be regularly followed (Fig.1). At baseline and week 16, a cardiac catheterization and MRI will assess changes in pulmonary hemodynamics and RV function.
  Other Names: BRD4 inhibitor

SUMMARY:
The main OBJECTIVE of this proposal is to extend the investigator's preclinical findings on the role of epigenetics and DNA damage and Bromodomain-Containing Protein 4 (BRD4) inhibition as a therapy for a devastating disease, pulmonary arterial hypertension (PAH).

There is strong evidence that BRD4 plays a key role in the pathological phenotype in PAH accounting for disease progression and that BRD4 inhibition can reverse PAH in several animal models. Intriguingly, coronary artery disease (CAD) and metabolic syndrome are more prevalent in PAH compared with the global population, suggesting a link between these diseases. Interestingly, BRD4 is also a trigger for calcification and remodeling processes and regulates transcription of lipoprotein and inflammatory factors, all of which are important in PAH and CAD. Apabetalone, an orally available BRD4 inhibitor, is now in a clinical development stage with a good safety profile.

At this stage, the investigators propose a pilot study to assess the feasibility of a Phase 2 clinical trial assessing apabetalone in the PAH population. The overall HYPOTHESIS is that BRD4 inhibition with apabetalone is a safe and effective therapy for PAH.

DETAILED DESCRIPTION:
In line with most pilot and safety studies, this is a two-centre (Quebec and Calgary) open-label trial. A 4-week pre-treatment phase will allow ensuring that patients are on stable doses of medication. Patients will be given doses of apabetalone 100mg BID for 16 weeks. Patients will be regularly followed. At baseline and week 16, a cardiac catheterization and MRI will assess changes in pulmonary hemodynamics and RV function.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-75 yrs) with PAH of idiopathic or hereditary origin, associated with connective tissue diseases, or anorexigen use.
2. Mean PA pressure ≥25mmHg, with pulmonary artery wedge pressure ≤15mmHg. In addition, subjects will be required meet the following hemodynamic criteria:

   1. PVR >480 dyn.s.cm-5
   2. Negative vasoreactivity test mandatory in idiopathic, heritable, and drug/toxin induced PAH (at baseline or during previous RHC).
3. World Health Organization functional class (WHO FC) II or III.
4. Appropriate stable therapy for PAH for ≥4 months before screening, including endothelin receptor antagonists (ERAs) other than bosentan and/or phosphodiesterase type 5 (PDE-5) inhibitors and/or prostanoids.
5. Two 6-min walk tests of 150-550m inclusive and within ±15% of each other (the latter being used as baseline value).
6. Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent.
7. Patients of childbearing potential must have a negative serum pregnancy test (β-hCG) within 72 hours prior to receiving the first dose of study treatment.
8. Patients must be postmenopausal, free from menses for >1 year, surgically sterilized, willing to use adequate contraception to prevent pregnancy, or agree to abstain from activities that could result in pregnancy, from enrollment through 3 months after the last dose of study treatment.

Exclusion Criteria:

1. PAH related to HIV infection, portal hypertension or congenital heart disease.
2. Pulmonary hypertension due to left heart disease (WHO PH group 2), lung disease and/or hypoxia (WHO PH group 3), chronic thromboembolic pulmonary hypertension (WHO PH group 4), or unclear multifactorial mechanisms (WHO PH group 5).
3. Known or suspected pulmonary veno-occlusive disease (PVOD).
4. Severe restrictive lung disease (Total Lung Capacity <60% predicted)
5. Severe obstructive lung disease (FEV1/FVC < 60% after a bronchodilator)
6. DLCO <40%
7. Systolic blood pressure <90 mmHg
8. Resting heart rate in the awake patient <50 BPM or >110 BPM
9. Clinically unstable right heart failure within the last 3 months or are WHO FC IV.
10. Received any investigational drug within 30 days of screening.
11. Body mass index (BMI) <18 or >40 kg/m2 at screening.
12. Patients must not be pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and for 3 months after the last dose of study treatment.
13. Cardiopulmonary rehabilitation program based on exercise (planned or started ≤12 weeks prior to Day 1).
14. Presence of ≥3 of the following risk factors for heart failure with preserved ejection fraction at screening:

    1. BMI >30 kg/m2.
    2. Diabetes mellitus of any type.
    3. Essential hypertension.
    4. Coronary artery disease, i.e., any of the following:

    i. History of stable angina ii. More than 50% stenosis in a coronary artery (by coronary angiography) iii. History of myocardial infarction iv. History of or planned coronary artery bypass grafting and/or coronary artery stenting.
15. A ventilation-perfusion lung scan or pulmonary angiography indicative of thromboembolic disease.
16. Evidence of organ dysfunction other than right heart failure, including:

    1. Creatinine clearance <45 ml/min (using the Cockroft-Gault formula).
    2. Serum AST or ALT >3 x ULN.
    3. Total bilirubin > 1.5 x ULN.
    4. Childs-Pugh class B-C liver cirrhosis.
    5. Hemoglobin <100 g/L.
    6. Absolute neutrophil count < 1,500/μL .
    7. Platelets < 150,000/μL .
17. Anticipated survival less than 1 year due to concomitant disease.
18. History of cancer in the past 5 years (except for low grade and fully resolved non-melanoma skin cancer).
19. Hypersensitivity to the components of apabetalone or any excipient of their formulations.

Forbidden concomitant therapy:

* Any investigational drug other than the study treatment.
* Based on in vitro data and clinical exposure data, apabetalone is considered unlikely to cause clinically significant drug interactions through inhibition or induction of cytochrome P450 enzyme activity. Nonetheless, as the contribution of metabolic clearance to total drug clearance in man is unknown, potent inhibitors (ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfanavir) or inducers (Phenytoin, rifampicin, carbamazepine and phenobarbitone, nevirapine, modafinil and St John's Wort) of CYP3A4 must not be used during this study for any patient receiving apabetalone to ensure patient safety. Moreover, bosentan has been associated with a 5-10% risk or reversible raised in LFTs. Although there is no evidence of increased risk of apabetalone-related increases in LFTs amongst bosentan users, the use of bosentan will be forbidden during this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Vascular Resistance (PVR), dyn·s·cm-5 | Baseline,and 16 weeks later
  Right heart catheterization: Measuring PVR is performed in a standardized manner in catheterization laboratories of the participating centres, according to recommendations. Printed copies of waveforms will be kept for monitoring visits and documentation of the accuracy of the pressures and calculations.

OTHER OUTCOMES:
Change in mean Pulmonary Artery Pressure (mPAP), mmHg | At screening and 16 weeks later
  The hemodynamic definition of pulmonary arterial hypertension (PAH) is a mean pulmonary artery pressure at rest greater than or equal to 25 mmHg in the presence of a pulmonary capillary wedge pressure less than or equal to 15 mmHg. These measurements can only be taken accurately during a right heart catheterization.
Change in cardiac output (L/min) | At screening and 16 weeks later
  Catheterization
Change in right atrial pressure (RAP), mmHg | At screening and 16 weeks later
  Catheterization
Change in mixed venous oxygen saturation (SvO2), % | At screening and 16 weeks later
  Catheterization
Change in the 6-min walk distance (6MWD), meters | Screening, Week 0 (baseline), Week 4, Week 8 and Week 16
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Change in WHO functional class | Screening, Week 0 (baseline), Week 4, Week 8, Week 16 and end of study
  There are four functional classes that are used to rate how ill PH patients are. Class I: No symptoms of pulmonary arterial hypertension with exercise or at rest. Class II: No symptoms at rest but uncomfortable and short of breath with normal activity such as climbing a flight of stairs, grocery shopping, or making the bed. Class III: May not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting. Class IV: Symptoms at rest and severe symptoms with any activity.
Change in plasma N-terminal pro-brain natriuretic peptide (NT-proBNP) concentration | Week 0 (baseline), Week 8, and Week 16
  To assess changes in inflammatory/calcification mediators (mRNA & serum proteins) of PAH patients with apabetalone treatment and demonstrate on-target beneficial effects, plasma (EDTA tubes) and whole blood (mRNA; PAXgene tubes) samples will be collected in subjects at visits 0 (baseline), 8 weeks, and 16 weeks. Blood draws at the 8 and 16 week visits should occur 4-6 hours post apabetalone dose to optimize capture of apabetalone's impact on gene expression (mRNA analysis). The plasma samples (EDTA tubes) will be processed and stored at -80°C until shipment on dry ice for future exploratory biomarker analysis relevant to lipid and inflammatory pathways. Whole blood samples (PAXgene tubes) will be stored at -20°C until shipment on dry ice to evaluate gene expression changes.
Change in Quality of life (QoL) using Emphasis-10 questionnaire | Week 0 (baseline), and Week 16
  The Emphasis-10 questionnaire is a short questionnaire for assessing HRQoL in pulmonary arterial hypertension. It has excellent measurement properties and is sensitive to differences in relevant clinical parameters.
Change in biomarker samples | Week 0 (baseline), Week 8, and Week 16
  circulating levels and transcription (messenger RNA) changes in whole blood of vascular calcification markers (alkaline phosphatase, osteoprotegerin), inflammation (C-reactive protein, fibrinogen, and inflammatory cytokines), complement, acute phase response, fibrogenesis and metabolism (adiponectin, ApoA-I, LDL-C and HDL-C)

CONTACTS AND LOCATIONS:
Overall Officials: Steeve Provencher, MD, MSc, Principal Investigator — IUCPQ-UL; Sébastien Bonnet, PhD, FAHA, Principal Investigator — IUCPQ-UL; Pascale Blais-Lecours, PhD, Study Director — IUCPQ-UL
Locations (2):
- Canada (2):
  - Peter Lougheed Center, Calgary, Alberta
  - IUCPQ-UL, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meloche J, Potus F, Vaillancourt M, Bourgeois A, Johnson I, Deschamps L, Chabot S, Ruffenach G, Henry S, Breuils-Bonnet S, Tremblay E, Nadeau V, Lambert C, Paradis R, Provencher S, Bonnet S. Bromodomain-Containing Protein 4: The Epigenetic Origin of Pulmonary Arterial Hypertension. Circ Res. 2015 Aug 28;117(6):525-35. doi: 10.1161/CIRCRESAHA.115.307004. Epub 2015 Jul 29. PMID 26224795
- [Background] Meloche J, Lampron MC, Nadeau V, Maltais M, Potus F, Lambert C, Tremblay E, Vitry G, Breuils-Bonnet S, Boucherat O, Charbonneau E, Provencher S, Paulin R, Bonnet S. Implication of Inflammation and Epigenetic Readers in Coronary Artery Remodeling in Patients With Pulmonary Arterial Hypertension. Arterioscler Thromb Vasc Biol. 2017 Aug;37(8):1513-1523. doi: 10.1161/ATVBAHA.117.309156. Epub 2017 May 4. PMID 28473439
- [Background] Paulin R, Michelakis ED. The metabolic theory of pulmonary arterial hypertension. Circ Res. 2014 Jun 20;115(1):148-64. doi: 10.1161/CIRCRESAHA.115.301130. PMID 24951764
- [Background] Zamanian RT, Hansmann G, Snook S, Lilienfeld D, Rappaport KM, Reaven GM, Rabinovitch M, Doyle RL. Insulin resistance in pulmonary arterial hypertension. Eur Respir J. 2009 Feb;33(2):318-24. doi: 10.1183/09031936.00000508. Epub 2008 Dec 1. PMID 19047320
- [Background] Ruffenach G, Chabot S, Tanguay VF, Courboulin A, Boucherat O, Potus F, Meloche J, Pflieger A, Breuils-Bonnet S, Nadeau V, Paradis R, Tremblay E, Girerd B, Hautefort A, Montani D, Fadel E, Dorfmuller P, Humbert M, Perros F, Paulin R, Provencher S, Bonnet S. Role for Runt-related Transcription Factor 2 in Proliferative and Calcified Vascular Lesions in Pulmonary Arterial Hypertension. Am J Respir Crit Care Med. 2016 Nov 15;194(10):1273-1285. doi: 10.1164/rccm.201512-2380OC. PMID 27149112
- [Background] Lehmann N, Erbel R, Mahabadi AA, Rauwolf M, Mohlenkamp S, Moebus S, Kalsch H, Budde T, Schmermund A, Stang A, Fuhrer-Sakel D, Weimar C, Roggenbuck U, Dragano N, Jockel KH; Heinz Nixdorf Recall Study Investigators. Value of Progression of Coronary Artery Calcification for Risk Prediction of Coronary and Cardiovascular Events: Result of the HNR Study (Heinz Nixdorf Recall). Circulation. 2018 Feb 13;137(7):665-679. doi: 10.1161/CIRCULATIONAHA.116.027034. Epub 2017 Nov 15. PMID 29142010
- [Background] Nicholls SJ, Puri R, Wolski K, Ballantyne CM, Barter PJ, Brewer HB, Kastelein JJ, Hu B, Uno K, Kataoka Y, Herrman JP, Merkely B, Borgman M, Nissen SE. Effect of the BET Protein Inhibitor, RVX-208, on Progression of Coronary Atherosclerosis: Results of the Phase 2b, Randomized, Double-Blind, Multicenter, ASSURE Trial. Am J Cardiovasc Drugs. 2016 Feb;16(1):55-65. doi: 10.1007/s40256-015-0146-z. PMID 26385396
- [Background] Vonk-Noordegraaf A, Haddad F, Chin KM, Forfia PR, Kawut SM, Lumens J, Naeije R, Newman J, Oudiz RJ, Provencher S, Torbicki A, Voelkel NF, Hassoun PM. Right heart adaptation to pulmonary arterial hypertension: physiology and pathobiology. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D22-33. doi: 10.1016/j.jacc.2013.10.027. PMID 24355638
- [Background] Bogaard HJ, Abe K, Vonk Noordegraaf A, Voelkel NF. The right ventricle under pressure: cellular and molecular mechanisms of right-heart failure in pulmonary hypertension. Chest. 2009 Mar;135(3):794-804. doi: 10.1378/chest.08-0492. PMID 19265089
- [Background] Lajoie AC, Lauziere G, Lega JC, Lacasse Y, Martin S, Simard S, Bonnet S, Provencher S. Combination therapy versus monotherapy for pulmonary arterial hypertension: a meta-analysis. Lancet Respir Med. 2016 Apr;4(4):291-305. doi: 10.1016/S2213-2600(16)00027-8. Epub 2016 Feb 27. PMID 26935844
- [Background] Humbert M, Lau EM, Montani D, Jais X, Sitbon O, Simonneau G. Advances in therapeutic interventions for patients with pulmonary arterial hypertension. Circulation. 2014 Dec 9;130(24):2189-208. doi: 10.1161/CIRCULATIONAHA.114.006974. No abstract available. PMID 25602947
- [Background] Humbert M, Sitbon O, Yaici A, Montani D, O'Callaghan DS, Jais X, Parent F, Savale L, Natali D, Gunther S, Chaouat A, Chabot F, Cordier JF, Habib G, Gressin V, Jing ZC, Souza R, Simonneau G; French Pulmonary Arterial Hypertension Network. Survival in incident and prevalent cohorts of patients with pulmonary arterial hypertension. Eur Respir J. 2010 Sep;36(3):549-55. doi: 10.1183/09031936.00057010. Epub 2010 Jun 18. PMID 20562126
- [Background] Humbert M, Sitbon O, Chaouat A, Bertocchi M, Habib G, Gressin V, Yaici A, Weitzenblum E, Cordier JF, Chabot F, Dromer C, Pison C, Reynaud-Gaubert M, Haloun A, Laurent M, Hachulla E, Cottin V, Degano B, Jais X, Montani D, Souza R, Simonneau G. Survival in patients with idiopathic, familial, and anorexigen-associated pulmonary arterial hypertension in the modern management era. Circulation. 2010 Jul 13;122(2):156-63. doi: 10.1161/CIRCULATIONAHA.109.911818. Epub 2010 Jun 28. PMID 20585011
- [Background] Benza RL, Gomberg-Maitland M, Miller DP, Frost A, Frantz RP, Foreman AJ, Badesch DB, McGoon MD. The REVEAL Registry risk score calculator in patients newly diagnosed with pulmonary arterial hypertension. Chest. 2012 Feb;141(2):354-362. doi: 10.1378/chest.11-0676. Epub 2011 Jun 16. PMID 21680644
- [Background] Benza RL, Miller DP, Gomberg-Maitland M, Frantz RP, Foreman AJ, Coffey CS, Frost A, Barst RJ, Badesch DB, Elliott CG, Liou TG, McGoon MD. Predicting survival in pulmonary arterial hypertension: insights from the Registry to Evaluate Early and Long-Term Pulmonary Arterial Hypertension Disease Management (REVEAL). Circulation. 2010 Jul 13;122(2):164-72. doi: 10.1161/CIRCULATIONAHA.109.898122. Epub 2010 Jun 28. PMID 20585012
- [Background] Escribano-Subias P, Blanco I, Lopez-Meseguer M, Lopez-Guarch CJ, Roman A, Morales P, Castillo-Palma MJ, Segovia J, Gomez-Sanchez MA, Barbera JA; REHAP investigators. Survival in pulmonary hypertension in Spain: insights from the Spanish registry. Eur Respir J. 2012 Sep;40(3):596-603. doi: 10.1183/09031936.00101211. Epub 2012 Feb 23. PMID 22362843
- [Background] Bonnet S, Michelakis ED, Porter CJ, Andrade-Navarro MA, Thebaud B, Bonnet S, Haromy A, Harry G, Moudgil R, McMurtry MS, Weir EK, Archer SL. An abnormal mitochondrial-hypoxia inducible factor-1alpha-Kv channel pathway disrupts oxygen sensing and triggers pulmonary arterial hypertension in fawn hooded rats: similarities to human pulmonary arterial hypertension. Circulation. 2006 Jun 6;113(22):2630-41. doi: 10.1161/CIRCULATIONAHA.105.609008. Epub 2006 May 30. PMID 16735674
- [Background] Paulin R, Courboulin A, Meloche J, Mainguy V, Dumas de la Roque E, Saksouk N, Cote J, Provencher S, Sussman MA, Bonnet S. Signal transducers and activators of transcription-3/pim1 axis plays a critical role in the pathogenesis of human pulmonary arterial hypertension. Circulation. 2011 Mar 22;123(11):1205-15. doi: 10.1161/CIRCULATIONAHA.110.963314. Epub 2011 Mar 7. PMID 21382889
- [Background] Guignabert C, Tu L, Le Hiress M, Ricard N, Sattler C, Seferian A, Huertas A, Humbert M, Montani D. Pathogenesis of pulmonary arterial hypertension: lessons from cancer. Eur Respir Rev. 2013 Dec;22(130):543-51. doi: 10.1183/09059180.00007513. PMID 24293470
- [Background] Leopold JA, Maron BA. Molecular Mechanisms of Pulmonary Vascular Remodeling in Pulmonary Arterial Hypertension. Int J Mol Sci. 2016 May 18;17(5):761. doi: 10.3390/ijms17050761. PMID 27213345
- [Background] Li MX, Jiang DQ, Wang Y, Chen QZ, Ma YJ, Yu SS, Wang Y. Signal Mechanisms of Vascular Remodeling in the Development of Pulmonary Arterial Hypertension. J Cardiovasc Pharmacol. 2016 Feb;67(2):182-90. doi: 10.1097/FJC.0000000000000328. PMID 26448276
- [Background] Meloche J, Pflieger A, Vaillancourt M, Paulin R, Potus F, Zervopoulos S, Graydon C, Courboulin A, Breuils-Bonnet S, Tremblay E, Couture C, Michelakis ED, Provencher S, Bonnet S. Role for DNA damage signaling in pulmonary arterial hypertension. Circulation. 2014 Feb 18;129(7):786-97. doi: 10.1161/CIRCULATIONAHA.113.006167. Epub 2013 Nov 22. PMID 24270264
- [Background] Li M, Vattulainen S, Aho J, Orcholski M, Rojas V, Yuan K, Helenius M, Taimen P, Myllykangas S, De Jesus Perez V, Koskenvuo JW, Alastalo TP. Loss of bone morphogenetic protein receptor 2 is associated with abnormal DNA repair in pulmonary arterial hypertension. Am J Respir Cell Mol Biol. 2014 Jun;50(6):1118-28. doi: 10.1165/rcmb.2013-0349OC. PMID 24433082
- [Background] Federici C, Drake KM, Rigelsky CM, McNelly LN, Meade SL, Comhair SA, Erzurum SC, Aldred MA. Increased Mutagen Sensitivity and DNA Damage in Pulmonary Arterial Hypertension. Am J Respir Crit Care Med. 2015 Jul 15;192(2):219-28. doi: 10.1164/rccm.201411-2128OC. PMID 25918951
- [Background] Rabinovitch M, Guignabert C, Humbert M, Nicolls MR. Inflammation and immunity in the pathogenesis of pulmonary arterial hypertension. Circ Res. 2014 Jun 20;115(1):165-75. doi: 10.1161/CIRCRESAHA.113.301141. PMID 24951765
- [Background] Happe CM, Szulcek R, Voelkel NF, Bogaard HJ. Reconciling paradigms of abnormal pulmonary blood flow and quasi-malignant cellular alterations in pulmonary arterial hypertension. Vascul Pharmacol. 2016 Aug;83:17-25. doi: 10.1016/j.vph.2016.01.004. Epub 2016 Jan 22. PMID 26804008
- [Background] Bonnet S, Rochefort G, Sutendra G, Archer SL, Haromy A, Webster L, Hashimoto K, Bonnet SN, Michelakis ED. The nuclear factor of activated T cells in pulmonary arterial hypertension can be therapeutically targeted. Proc Natl Acad Sci U S A. 2007 Jul 3;104(27):11418-23. doi: 10.1073/pnas.0610467104. Epub 2007 Jun 27. PMID 17596340
- [Background] Courboulin A, Paulin R, Giguere NJ, Saksouk N, Perreault T, Meloche J, Paquet ER, Biardel S, Provencher S, Cote J, Simard MJ, Bonnet S. Role for miR-204 in human pulmonary arterial hypertension. J Exp Med. 2011 Mar 14;208(3):535-48. doi: 10.1084/jem.20101812. Epub 2011 Feb 14. PMID 21321078
- [Background] Bonnet S, Provencher S, Guignabert C, Perros F, Boucherat O, Schermuly RT, Hassoun PM, Rabinovitch M, Nicolls MR, Humbert M. Translating Research into Improved Patient Care in Pulmonary Arterial Hypertension. Am J Respir Crit Care Med. 2017 Mar 1;195(5):583-595. doi: 10.1164/rccm.201607-1515PP. No abstract available. PMID 27649290
- [Background] Lamoureux F, Baud'huin M, Rodriguez Calleja L, Jacques C, Berreur M, Redini F, Lecanda F, Bradner JE, Heymann D, Ory B. Selective inhibition of BET bromodomain epigenetic signalling interferes with the bone-associated tumour vicious cycle. Nat Commun. 2014 Mar 19;5:3511. doi: 10.1038/ncomms4511. PMID 24646477
- [Background] Wyce A, Ganji G, Smitheman KN, Chung CW, Korenchuk S, Bai Y, Barbash O, Le B, Craggs PD, McCabe MT, Kennedy-Wilson KM, Sanchez LV, Gosmini RL, Parr N, McHugh CF, Dhanak D, Prinjha RK, Auger KR, Tummino PJ. BET inhibition silences expression of MYCN and BCL2 and induces cytotoxicity in neuroblastoma tumor models. PLoS One. 2013 Aug 23;8(8):e72967. doi: 10.1371/journal.pone.0072967. eCollection 2013. PMID 24009722
- [Background] Baratta MG, Schinzel AC, Zwang Y, Bandopadhayay P, Bowman-Colin C, Kutt J, Curtis J, Piao H, Wong LC, Kung AL, Beroukhim R, Bradner JE, Drapkin R, Hahn WC, Liu JF, Livingston DM. An in-tumor genetic screen reveals that the BET bromodomain protein, BRD4, is a potential therapeutic target in ovarian carcinoma. Proc Natl Acad Sci U S A. 2015 Jan 6;112(1):232-7. doi: 10.1073/pnas.1422165112. Epub 2014 Dec 22. PMID 25535366
- [Background] Tolani B, Gopalakrishnan R, Punj V, Matta H, Chaudhary PM. Targeting Myc in KSHV-associated primary effusion lymphoma with BET bromodomain inhibitors. Oncogene. 2014 May 29;33(22):2928-37. doi: 10.1038/onc.2013.242. Epub 2013 Jun 24. PMID 23792448
- [Background] Gallagher SJ, Mijatov B, Gunatilake D, Tiffen JC, Gowrishankar K, Jin L, Pupo GM, Cullinane C, Prinjha RK, Smithers N, McArthur GA, Rizos H, Hersey P. The epigenetic regulator I-BET151 induces BIM-dependent apoptosis and cell cycle arrest of human melanoma cells. J Invest Dermatol. 2014 Nov;134(11):2795-2805. doi: 10.1038/jid.2014.243. Epub 2014 Jun 6. PMID 24906137
- [Background] Belkina AC, Denis GV. BET domain co-regulators in obesity, inflammation and cancer. Nat Rev Cancer. 2012 Jun 22;12(7):465-77. doi: 10.1038/nrc3256. PMID 22722403
- [Background] Segura MF, Fontanals-Cirera B, Gaziel-Sovran A, Guijarro MV, Hanniford D, Zhang G, Gonzalez-Gomez P, Morante M, Jubierre L, Zhang W, Darvishian F, Ohlmeyer M, Osman I, Zhou MM, Hernando E. BRD4 sustains melanoma proliferation and represents a new target for epigenetic therapy. Cancer Res. 2013 Oct 15;73(20):6264-76. doi: 10.1158/0008-5472.CAN-13-0122-T. Epub 2013 Aug 15. PMID 23950209
- [Background] Rahman S, Sowa ME, Ottinger M, Smith JA, Shi Y, Harper JW, Howley PM. The Brd4 extraterminal domain confers transcription activation independent of pTEFb by recruiting multiple proteins, including NSD3. Mol Cell Biol. 2011 Jul;31(13):2641-52. doi: 10.1128/MCB.01341-10. Epub 2011 May 9. PMID 21555454
- [Background] Kanno T, Kanno Y, LeRoy G, Campos E, Sun HW, Brooks SR, Vahedi G, Heightman TD, Garcia BA, Reinberg D, Siebenlist U, O'Shea JJ, Ozato K. BRD4 assists elongation of both coding and enhancer RNAs by interacting with acetylated histones. Nat Struct Mol Biol. 2014 Dec;21(12):1047-57. doi: 10.1038/nsmb.2912. Epub 2014 Nov 10. PMID 25383670
- [Background] Devaiah BN, Lewis BA, Cherman N, Hewitt MC, Albrecht BK, Robey PG, Ozato K, Sims RJ 3rd, Singer DS. BRD4 is an atypical kinase that phosphorylates serine2 of the RNA polymerase II carboxy-terminal domain. Proc Natl Acad Sci U S A. 2012 May 1;109(18):6927-32. doi: 10.1073/pnas.1120422109. Epub 2012 Apr 16. PMID 22509028
- [Background] Berthon C, Raffoux E, Thomas X, Vey N, Gomez-Roca C, Yee K, Taussig DC, Rezai K, Roumier C, Herait P, Kahatt C, Quesnel B, Michallet M, Recher C, Lokiec F, Preudhomme C, Dombret H. Bromodomain inhibitor OTX015 in patients with acute leukaemia: a dose-escalation, phase 1 study. Lancet Haematol. 2016 Apr;3(4):e186-95. doi: 10.1016/S2352-3026(15)00247-1. Epub 2016 Mar 18. PMID 27063977
- [Background] Amorim S, Stathis A, Gleeson M, Iyengar S, Magarotto V, Leleu X, Morschhauser F, Karlin L, Broussais F, Rezai K, Herait P, Kahatt C, Lokiec F, Salles G, Facon T, Palumbo A, Cunningham D, Zucca E, Thieblemont C. Bromodomain inhibitor OTX015 in patients with lymphoma or multiple myeloma: a dose-escalation, open-label, pharmacokinetic, phase 1 study. Lancet Haematol. 2016 Apr;3(4):e196-204. doi: 10.1016/S2352-3026(16)00021-1. Epub 2016 Mar 18. PMID 27063978
- [Background] Belkina AC, Nikolajczyk BS, Denis GV. BET protein function is required for inflammation: Brd2 genetic disruption and BET inhibitor JQ1 impair mouse macrophage inflammatory responses. J Immunol. 2013 Apr 1;190(7):3670-8. doi: 10.4049/jimmunol.1202838. Epub 2013 Feb 18. PMID 23420887
- [Background] Brown JD, Lin CY, Duan Q, Griffin G, Federation A, Paranal RM, Bair S, Newton G, Lichtman A, Kung A, Yang T, Wang H, Luscinskas FW, Croce K, Bradner JE, Plutzky J. NF-kappaB directs dynamic super enhancer formation in inflammation and atherogenesis. Mol Cell. 2014 Oct 23;56(2):219-231. doi: 10.1016/j.molcel.2014.08.024. Epub 2014 Sep 25. PMID 25263595
- [Background] Khan YM, Kirkham P, Barnes PJ, Adcock IM. Brd4 is essential for IL-1beta-induced inflammation in human airway epithelial cells. PLoS One. 2014 Apr 23;9(4):e95051. doi: 10.1371/journal.pone.0095051. eCollection 2014. PMID 24759736
- [Background] Mercer JR, Cheng KK, Figg N, Gorenne I, Mahmoudi M, Griffin J, Vidal-Puig A, Logan A, Murphy MP, Bennett M. DNA damage links mitochondrial dysfunction to atherosclerosis and the metabolic syndrome. Circ Res. 2010 Oct 15;107(8):1021-31. doi: 10.1161/CIRCRESAHA.110.218966. Epub 2010 Aug 12. PMID 20705925
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Tang X, Peng R, Phillips JE, Deguzman J, Ren Y, Apparsundaram S, Luo Q, Bauer CM, Fuentes ME, DeMartino JA, Tyagi G, Garrido R, Hogaboam CM, Denton CP, Holmes AM, Kitson C, Stevenson CS, Budd DC. Assessment of Brd4 inhibition in idiopathic pulmonary fibrosis lung fibroblasts and in vivo models of lung fibrosis. Am J Pathol. 2013 Aug;183(2):470-9. doi: 10.1016/j.ajpath.2013.04.020. Epub 2013 Jun 10. PMID 23759512
- [Background] Zou Z, Huang B, Wu X, Zhang H, Qi J, Bradner J, Nair S, Chen LF. Brd4 maintains constitutively active NF-kappaB in cancer cells by binding to acetylated RelA. Oncogene. 2014 May 1;33(18):2395-404. doi: 10.1038/onc.2013.179. Epub 2013 May 20. PMID 23686307
- [Background] Stanlie A, Yousif AS, Akiyama H, Honjo T, Begum NA. Chromatin reader Brd4 functions in Ig class switching as a repair complex adaptor of nonhomologous end-joining. Mol Cell. 2014 Jul 3;55(1):97-110. doi: 10.1016/j.molcel.2014.05.018. Epub 2014 Jun 19. PMID 24954901
- [Background] Lee DH, Qi J, Bradner JE, Said JW, Doan NB, Forscher C, Yang H, Koeffler HP. Synergistic effect of JQ1 and rapamycin for treatment of human osteosarcoma. Int J Cancer. 2015 May 1;136(9):2055-64. doi: 10.1002/ijc.29269. Epub 2014 Oct 30. PMID 25307878
- [Background] Gilham D, Tsujikawa L, Wasiak S, et al. Apabetalone Downregulates Factors That Promote Vascular Calcification and Contribute to Cardiovascular Events. Circulation. 2017;136:A-15906.
- [Background] Hill BG, Benavides GA, Lancaster JR Jr, Ballinger S, Dell'Italia L, Jianhua Z, Darley-Usmar VM. Integration of cellular bioenergetics with mitochondrial quality control and autophagy. Biol Chem. 2012 Dec;393(12):1485-1512. doi: 10.1515/hsz-2012-0198. PMID 23092819
- [Background] Hautefort A, Girerd B, Montani D, Cohen-Kaminsky S, Price L, Lambrecht BN, Humbert M, Perros F. T-helper 17 cell polarization in pulmonary arterial hypertension. Chest. 2015 Jun;147(6):1610-1620. doi: 10.1378/chest.14-1678. PMID 25429518
- [Background] Mele DA, Salmeron A, Ghosh S, Huang HR, Bryant BM, Lora JM. BET bromodomain inhibition suppresses TH17-mediated pathology. J Exp Med. 2013 Oct 21;210(11):2181-90. doi: 10.1084/jem.20130376. Epub 2013 Oct 7. PMID 24101376
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] McLaughlin VV, Badesch DB, Delcroix M, Fleming TR, Gaine SP, Galie N, Gibbs JSR, Kim NH, Oudiz RJ, Peacock A, Provencher S, Sitbon O, Tapson VF, Seeger W. End points and clinical trial design in pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S97-S107. doi: 10.1016/j.jacc.2009.04.007. PMID 19555863
- [Background] Mainguy V, Provencher S, Maltais F, Malenfant S, Saey D. Assessment of daily life physical activities in pulmonary arterial hypertension. PLoS One. 2011;6(11):e27993. doi: 10.1371/journal.pone.0027993. Epub 2011 Nov 16. PMID 22110770
- [Background] Johnson SR, Swiston JR, Granton JT. Prognostic factors for survival in scleroderma associated pulmonary arterial hypertension. J Rheumatol. 2008 Aug;35(8):1584-90. Epub 2008 Jul 1. PMID 18597400
- [Background] Swiston JR, Johnson SR, Granton JT. Factors that prognosticate mortality in idiopathic pulmonary arterial hypertension: a systematic review of the literature. Respir Med. 2010 Nov;104(11):1588-607. doi: 10.1016/j.rmed.2010.08.003. PMID 20810261
- [Background] Souza R, Jardim C, Carvalho C, Rubenfeld G. The role of NT-proBNP as a prognostic marker in pulmonary hypertension. Chest. 2006 Nov;130(5):1627; author reply 1627-8. doi: 10.1378/chest.130.5.1627. No abstract available. PMID 17099052
- [Background] Gan CT, McCann GP, Marcus JT, van Wolferen SA, Twisk JW, Boonstra A, Postmus PE, Vonk-Noordegraaf A. NT-proBNP reflects right ventricular structure and function in pulmonary hypertension. Eur Respir J. 2006 Dec;28(6):1190-4. doi: 10.1183/09031936.00016006. Epub 2006 Sep 13. PMID 16971413
- [Background] Chin KM, Channick RN, Kim NH, Rubin LJ. Central venous blood oxygen saturation monitoring in patients with chronic pulmonary arterial hypertension treated with continuous IV epoprostenol: correlation with measurements of hemodynamics and plasma brain natriuretic peptide levels. Chest. 2007 Sep;132(3):786-92. doi: 10.1378/chest.07-0694. Epub 2007 Jul 23. PMID 17646224
- [Background] Giannakoulas G, Dimopoulos K, Bolger AP, Tay EL, Inuzuka R, Bedard E, Davos C, Swan L, Gatzoulis MA. Usefulness of natriuretic Peptide levels to predict mortality in adults with congenital heart disease. Am J Cardiol. 2010 Mar 15;105(6):869-73. doi: 10.1016/j.amjcard.2009.11.041. PMID 20211335
- [Background] Nagaya N, Nishikimi T, Uematsu M, Satoh T, Kyotani S, Sakamaki F, Kakishita M, Fukushima K, Okano Y, Nakanishi N, Miyatake K, Kangawa K. [Plasma brain natriuretic peptide as a prognostic indicator in patients with primary pulmonary hypertension]. J Cardiol. 2001 Feb;37(2):110-1. Japanese. PMID 11255693
- [Background] Rival G, Lacasse Y, Martin S, Bonnet S, Provencher S. Effect of pulmonary arterial hypertension-specific therapies on health-related quality of life: a systematic review. Chest. 2014 Sep;146(3):686-708. doi: 10.1378/chest.13-2634. PMID 24626791
- [Background] Hoeper MM, Bogaard HJ, Condliffe R, Frantz R, Khanna D, Kurzyna M, Langleben D, Manes A, Satoh T, Torres F, Wilkins MR, Badesch DB. Definitions and diagnosis of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D42-50. doi: 10.1016/j.jacc.2013.10.032. PMID 24355641
- [Background] Simonneau G, Gatzoulis MA, Adatia I, Celermajer D, Denton C, Ghofrani A, Gomez Sanchez MA, Krishna Kumar R, Landzberg M, Machado RF, Olschewski H, Robbins IM, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D34-41. doi: 10.1016/j.jacc.2013.10.029. PMID 24355639
- [Background] Boxt LM, Katz J, Kolb T, Czegledy FP, Barst RJ. Direct quantitation of right and left ventricular volumes with nuclear magnetic resonance imaging in patients with primary pulmonary hypertension. J Am Coll Cardiol. 1992 Jun;19(7):1508-15. doi: 10.1016/0735-1097(92)90611-p. PMID 1593046
- [Background] Katz J, Whang J, Boxt LM, Barst RJ. Estimation of right ventricular mass in normal subjects and in patients with primary pulmonary hypertension by nuclear magnetic resonance imaging. J Am Coll Cardiol. 1993 May;21(6):1475-81. doi: 10.1016/0735-1097(93)90327-w. PMID 8473659
- [Background] Lorenz CH, Walker ES, Morgan VL, Klein SS, Graham TP Jr. Normal human right and left ventricular mass, systolic function, and gender differences by cine magnetic resonance imaging. J Cardiovasc Magn Reson. 1999;1(1):7-21. doi: 10.3109/10976649909080829. PMID 11550343
- [Background] Grothues F, Moon JC, Bellenger NG, Smith GS, Klein HU, Pennell DJ. Interstudy reproducibility of right ventricular volumes, function, and mass with cardiovascular magnetic resonance. Am Heart J. 2004 Feb;147(2):218-23. doi: 10.1016/j.ahj.2003.10.005. PMID 14760316
- [Background] Semelka RC, Tomei E, Wagner S, Mayo J, Caputo G, O'Sullivan M, Parmley WW, Chatterjee K, Wolfe C, Higgins CB. Interstudy reproducibility of dimensional and functional measurements between cine magnetic resonance studies in the morphologically abnormal left ventricle. Am Heart J. 1990 Jun;119(6):1367-73. doi: 10.1016/s0002-8703(05)80187-5. PMID 2141222
- [Background] Semelka RC, Tomei E, Wagner S, Mayo J, Kondo C, Suzuki J, Caputo GR, Higgins CB. Normal left ventricular dimensions and function: interstudy reproducibility of measurements with cine MR imaging. Radiology. 1990 Mar;174(3 Pt 1):763-8. doi: 10.1148/radiology.174.3.2305059.
- [Background] Galie N, Manes A, Negro L, Palazzini M, Bacchi-Reggiani ML, Branzi A. A meta-analysis of randomized controlled trials in pulmonary arterial hypertension. Eur Heart J. 2009 Feb;30(4):394-403. doi: 10.1093/eurheartj/ehp022. Epub 2009 Jan 20. PMID 19155250
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] McKenna SP, Doughty N, Meads DM, Doward LC, Pepke-Zaba J. The Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR): a measure of health-related quality of life and quality of life for patients with pulmonary hypertension. Qual Life Res. 2006 Feb;15(1):103-15. doi: 10.1007/s11136-005-3513-4. PMID 16411035
- [Background] Taylor GJ, Wainwright P. Open label extension studies: research or marketing? BMJ. 2005 Sep 10;331(7516):572-4. doi: 10.1136/bmj.331.7516.572. PMID 16150772
- [Background] Micetich KC. The ethical problems of the open label extension study. Camb Q Healthc Ethics. 1996 Summer;5(3):410-4. doi: 10.1017/s0963180100007210. No abstract available. PMID 8862827
- [Background] Yorke J, Corris P, Gaine S, Gibbs JS, Kiely DG, Harries C, Pollock V, Armstrong I. emPHasis-10: development of a health-related quality of life measure in pulmonary hypertension. Eur Respir J. 2014 Apr;43(4):1106-13. doi: 10.1183/09031936.00127113. Epub 2013 Nov 14. PMID 24232702
- [Background] Yorke J, Deaton C, Campbell M, McGowen L, Sephton P, Kiely DG, Armstrong I. Symptom severity and its effect on health-related quality of life over time in patients with pulmonary hypertension: a multisite longitudinal cohort study. BMJ Open Respir Res. 2018 Mar 1;5(1):e000263. doi: 10.1136/bmjresp-2017-000263. eCollection 2018. PMID 29531745
- [Background] Favoccia C, Kempny A, Yorke J, Armstrong I, Price LC, McCabe C, Harries C, Wort SJ, Dimopoulos K. EmPHasis-10 score for the assessment of quality of life in various types of pulmonary hypertension and its relation to outcome. Eur J Prev Cardiol. 2019 Aug;26(12):1338-1340. doi: 10.1177/2047487318819161. Epub 2018 Dec 19. No abstract available. PMID 30567456
- [Derived] Provencher S, Potus F, Blais-Lecours P, Bernard S, Martineau S, Breuils-Bonnet S, Weatherald J, Sweeney M, Kulikowski E, Boucherat O, Bonnet S. BET Protein Inhibition for Pulmonary Arterial Hypertension: A Pilot Clinical Trial. Am J Respir Crit Care Med. 2022 Jun 1;205(11):1357-1360. doi: 10.1164/rccm.202109-2182LE. No abstract available. PMID 35289736